CLINICAL TRIAL: NCT04800796
Title: Evaluation From Didactic and Structural Transfer of Standard Operating Procedures in Anesthesiology
Brief Title: Transfer of Standard Operating Procedures in Anesthesiology
Acronym: QUALI-II
Status: Completed | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Marc Kriege, MD, Principal Investigator, Johannes Gutenberg University Mainz
Other Study IDs: JohannesGUQ
Record Dates: First submitted 2021-03-09; First posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Patient Safety
MeSH Terms: interventions — Audiovisual Aids

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention Group: Intervention Group with audiovisually blended learning concept
  Interventions: Other: Audiovisual
- Standard group: Standard Group receiving the Standard operating procedures via E-Mail and Confirmation when reading.

INTERVENTIONS:
Other: Audiovisual — Receive blended learning before and reading the Standard operating procedure
  Groups: Intervention Group

SUMMARY:
Patients safety and high Quality Performance built up the centre of anesthesiology. Standard operating procedures based on the Helsinki declaration may help to increase the Patient safety and decreased adverse Events or complications.

DETAILED DESCRIPTION:
The Primary endpoint is the comparison of a Intervention Group with audiovisually blended learning concept and a Standard Group receiving the Standard operating procedures via E-Mail and Confirmation when reading.

ELIGIBILITY:
Inclusion:

* anesthesia residents
* anesthesia consultants

Exclusion:

* nurses
* students

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: anesthesia physicians who participating in a Scenario training
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-07 (Actual)

PRIMARY OUTCOMES:
Rate of SOP deviations | 12 minutes after start scenario
  SOP deviations during scenario training

CONTACTS AND LOCATIONS:
Overall Officials: Marc Kriege, MD, PhD, Principal Investigator — University JG, Mainz
Locations (1):
- Department of Anesthesiology,Prof. C. Werner, Universitätsmedizin of the JG University, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No